CLINICAL TRIAL: NCT04877899
Title: Mazankowski - Echo Go Discovery Protocol Retrospective LVEF/GLS Comparison
Brief Title: Mazankowski Alberta Heart Institute (MAHI) EchoGo Discovery 1 Protocol
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ultromics Ltd (Industry)
Collaborators: Mazankowski Alberta Heart Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: COL-04
Record Dates: First submitted 2021-04-22; First posted 2021-05-07 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Cardiotoxicity; Cancer
MeSH Terms: conditions — Cardiotoxicity; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: EchoGo — EchoGo Core is a stand-alone software application. Echocardiograms should be acquired under the supervision of a physician and standard clinical protocols which includes focused apical 2, 3 and 4 chamber views. The results contain calculated measurements that will be returned to the interpreting physician. These results are intended as an additional input to standard diagnostic pathways and should only be used by a board-certified cardiologist/physician.
  EchoGo Core is intended to be used for the quantification and reporting of results of cardiovascular function to support physician diagnosis. EchoGo Core is indicated for use in adult populations.

SUMMARY:
This study aims to compare conventionally acquired Left Ventricle Ejection Fraction (LVEF) and Global Longitudinal Strain (GLS) data to Artificial Intelligence (AI) driven automated processing of 2 dimensional contrast and 2 dimensional non-contrast resting transthoracic echocardiograms for application in the assessment of patients undergoing chemotherapy with cardiotoxic drugs. This is a single-centre retrospective study which utilizes echocardiographic DICOM image and meta-data datasets received from a Canadian site. Data processed using the AI driven automated processing will be compared to conventionally acquired LVEF and GLS measurements and results will be analysed to determine accuracy and precision.

ELIGIBILITY:
Inclusion Criteria:

* Normal EF and no regional wall motion abnormalities prior to starting chemotherapy treatment.
* Follow-up EF measurements available for at least 1 year during the treatment period.
* Follow-up EF measurements for at least 1 year during the treatment period.

Exclusion Criteria:

* Age < 18 years
* Inadequate image quality (as determined by the Ultromics Operators Quality Control process)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Data included for analysis in this study will be retrospective data from male and female patients aged 18 years or above who received an echocardiogram for baseline and follow-up of cardiotoxic agent management, who agreed to participate in the echocardiography registry of the MAHI, and who have already provided a written consent that their anonymized imaging data can be used to advance echocardiographic assessment of LV function.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Compare the performance of automated EF and GLS measurements in resting transthoracic echocardiograms against conventional measurement acquisition. | Baseline
  Measurements shall be compared using bias and 95% confidence intervals on bias. Regression coefficients and comparative statistics will be employed for this objective.
Compare the performance of automated EF and GLS measurements in resting transthoracic echocardiograms against conventional measurement acquisition. | Follow up (up to 1 year)
  Measurements shall be compared using bias and 95% confidence intervals on bias. Regression coefficients and comparative statistics will be employed for this objective.
Compare the performance of automated EF and GLS measurements in resting transthoracic echocardiograms with and without the application of contrast agents. | Baseline
  Measurements will be assessed using bias and 95% confidence internals on bias. Regression coefficients, comparative statistics and equivalence testing might also be employed as a comparison measure for this objective.
Compare the performance of automated EF and GLS measurements in resting transthoracic echocardiograms with and without the application of contrast agents. | Follow up (up to 1 year)
  Measurements will be assessed using bias and 95% confidence internals on bias. Regression coefficients, comparative statistics and equivalence testing might also be employed as a comparison measure for this objective.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Becher, Principal Investigator — Mazankowski Alberta Heart Institute
Locations (1):
- Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada